CLINICAL TRIAL: NCT05542615
Title: Evaluation of Prolonged-release Pirfenidone in Patients With Viral C Hepatitis, With Sustained Viral Response and Advanced Residual Liver Fibrosis. Potential Role of Epigenetics to Understand Therapeutic Changes (MINERVA).
Brief Title: Prolonged Release Pirfenidone for Advanced Residual Liver Fibrosis (MINERVA).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Central Militar (Other Government)
Responsible Party: Principal Investigator, Juan Armendáriz-Borunda, PhD, FAASLD, Director of Institute of Molecular Biology in Medicine, University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINERVA
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Liver Cirrhosis; Hepatitis C, Chronic; Epigenetic Disorder
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: This will be a real-life, open-label, proof of concept trial to assess the safety and efficacy of two daily doses of pirfenidone (KitosCell® LP), in patients with compensated liver cirrhosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental): Sixty patients with chronic Viral C hepatitis, who have been treated with direct-acting antivirals, with a sustained viral response and who still have advanced fibrosis (F3-F4).
  Interventions: Drug: Prolonged-Release Pirfenidone

INTERVENTIONS:
Drug: Prolonged-Release Pirfenidone — 1200 mg / day of Pirfenidone (KitosCell® LP)

SUMMARY:
Prolonged-Release Pirfenidone (PR-PFD) is an anti-fibrogenic and anti-inflammatory molecule used for the treatment of idiopathic pulmonary fibrosis (approved by FDA) and liver fibrosis (approved in Mexico by COFEPRIS). PFD effects are mediated in part through inhibition of TGFβ, TNFα, IL-1 and IL-6, along with NFκB activation down-regulation causing reduced TNFα and IFNγ levels.

The aim of this protocol is to know if the epigenetic factors induced by PR-PFD have a regulatory role to understand the progression variants in liver fibrosis in a group of patients with viral hepatitis C, with a history of sustained viral response and advanced residual liver fibrosis. To assess the safety and efficacy of two daily doses of pirfenidone (KitosCell® LP), in patients with compensated liver cirrhosis.

DETAILED DESCRIPTION:
Design: Observational clinical study, in an open population, of 12 months duration. Sixty patients with chronic Viral C hepatitis, who have been treated with direct-acting antivirals, with a sustained viral response and who still have advanced fibrosis (F3-F4).

Aim: to know if the epigenetic factors induced by PR-PFD have a regulatory role to understand the progression variants in liver fibrosis in a group of patients with viral hepatitis C, with a history of sustained viral response and advanced residual liver fibrosis. To assess the safety and efficacy of two daily doses of pirfenidone (KitosCell® LP), in patients with compensated liver cirrhosis.

Dosage: 1200 mg / day of Pirfenidone (KitosCell® LP) Variables to Analyze: Reduction of fibrosis and evaluation of epigenetic changes in the expression of various genes: PPARγ, PPARδ, PPARα, TGFβ1, Col1A1 and PDGFα. Additionally, changes in the expression levels of miR-122, miR192, miR-200a / b, miR-34a, miR-16, miR-21 and miR-181b will be evaluated, as well as changes in the transcriptome in ccfRNA.

Ethical considerations: The study will be conducted in accordance with the Declaration of Helsinki and the E6 Good Clinical Practice Standards International Conference on Harmonization (ICH).

Statistical Data Analysis: Descriptive statistics will be used and according to analytical statistical requirements that include parametric or non-parametric tests. The value of p <0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of Chronic Viral Hepatitis C, of all genotypes, demonstrated with previous studies (positive viral load).
2. History of treatment with direct acting antivirals (AAD).
3. Demonstration of negative viral load at least 6 months after completing treatment with AAD, considered as sustained viral response (SVR).
4. Fibrotest and / or Liver Elastography test with advanced liver fibrosis scores (F3-F4).
5. Verification of advanced liver fibrosis in a liver biopsy.
6. Patients with Child Pugh functional class A or B and in stable clinical conditions (without active variceal hemorrhage, ascites or refractory encephalopathy) with consumption of drugs at stable doses in at least 30 days.
7. Laboratory tests that confirm her condition and functional class, with results that, in the opinion of the main researcher, do not put the patient at risk:

   * Complete blood count, with hemoglobin values ≥ 10 g / dL, leukocytes ≥ 3,000 mL, platelets ≥ 50,000 mL
   * Creatinine <1.8 mg / dL

Exclusion Criteria:

1. Child Pugh functional class C (≥ 10 points)
2. Pregnancy and lactation.
3. History of known allergy or hypersensitivity to PFD.
4. Having participated in another clinical study in the 60 days prior to the start of this one.
5. Hospitalization within 30 days prior to the start of administration of the medication.
6. Co-existing liver pathology: alcohol cirrhosis, hemochromatosis, Wilson's disease, α-1-antitrypsin deficiency, amyloidosis, autoimmune hepatitis, and Primary Biliary Cholangitis).
7. Concomitant systemic infection including viral hepatitis B, HIV, as well as respiratory infections, urinary, digestive, cellulite, etc.
8. Serious concomitant conditions such as Heart Failure, Respiratory Failure and Chronic Kidney Failure.
9. Malignant neoplasms including hepatocellular carcinoma. Patients with basal cell carcinoma or those with malignancies with more than 5 years of inactivity may be considered for the study.
10. Decompensated diabetes mellitus (defined as that with fasting blood glucose values greater than 175 mg / dL and / or glycated hemoglobin greater than 8%).
11. Uncontrolled hypertension despite medications (defined as systolic values ≥ 150 and diastolic values ≥ 100 mmHg).
12. Patients with active alcohol intake in the last 6 months.
13. Use of drugs known as concomitant hepatoprotectors (ursodexosicolic acid, s-adenosyl-methionine, silymarin, among others).
14. Patients with treatment of CYP1A2 inhibitor drugs or other CYP isoenzymes such as: fluvoxamine, amiodarone, fluconazole, chloramphenicol, fluoxentine, paroxentine, ciprofloxacin, rifampin or propafenone, or other medicinal products that, in the opinion of the main investigator, may interfere with the study.
15. Any other clinical condition that in the opinion of the main investigator could compromise the safety and well-being of the patient or jeopardize the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Liver biopsy | 12 months
  Reduction of one unit in the METAVIR histological scale (F0-F4)
Elastography | 12 months
  ≥30% reduction in the final Pascal score, compared to baseline.

SECONDARY OUTCOMES:
Changes in the degree of methylation | 12 months
  of the following genes PPARγ, PPARζ, PPARα, TGFβ1, Col1A1 and PDGFα in ccfDNA in DNA obtained by liver biopsy.
Changes in expression levels of miRNA's | 12 months
  Changes in expression levels of miR-122, miR192, miR-200a / b, miR-221/222, miR-34a, miR-16, miR-21, and miR-181b.
Transcriptome measurement in ccfRNA | 12 months
  Changes in transcriptome measurement in ccfRNA
Albumin and liver enzyme values | 12 months
  Albumin and liver enzyme values

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Institute for Molecular Biology in Medicine and Gene Therapy, CUCS, UdeG, Guadalajara, Jalisco
  - Hospital Central Militar, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerda-Reyes E, de la Rosa-Bibiano R, Sandoval-Rodriguez A, Rosas-Campos R, Torre A, Cornejo-Hernandez S, Escutia-Gutierrez R, Vazquez-Esqueda A, Gutierrez-Cuevas J, Gutierrez-Atemis A, Amezquita-Perez S, Poo JL, Garrido-Sanchez GA, Bastida-Alquicira J, Saldana-Rivera E, Lozano-Trenado LM, Ramon-Aguilar J, Madrigal JA, Armendariz-Borunda J. HCV patients with residual fibrosis after DAA treatment re-establish their epigenetic signature after prolonged-release pirfenidone: MINERVA study. Clin Epigenetics. 2025 Oct 3;17(1):157. doi: 10.1186/s13148-025-01969-y. PMID 41044745